CLINICAL TRIAL: NCT06635980
Title: A Randomized Phase II Trial of Hypofractionated Radiotherapy for Non-Metastatic Breast Cancer Before or After Breast Surgery for Different Breast Cancer Risk Groups
Brief Title: Hypofractionated Radiotherapy Before or After Breast Surgery for Treatment of Patients With Non-Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROA2234; NCI-2024-08356 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-009070 (Other: Mayo Clinic Institutional Review Board); GMROA2234 (Other: Mayo Clinic Radiation Oncology)
Record Dates: First submitted 2024-10-09; First posted 2024-10-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Specimen Handling; Mastectomy, Segmental; Drug Therapy; Radiation Dose Hypofractionation; Radiation; Magnetic Resonance Spectroscopy; Tissue Banks; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Preoperative radiation therapy + surgery) (Experimental): Patients undergo SOC chemotherapy followed by breast hypofractionated radiotherapy QD for a total of 5 fractions. Patients then undergo SOC breast surgery 10 weeks after radiation treatment. Patients also undergo CT, MRI, PET, CEDM, and/or breast US throughout the study. Additionally, patients undergo a breast biopsy and may undergo optional blood sample collection and tissue collection on study.
  Interventions: Procedure: Biopsy of Breast; Procedure: Biospecimen Collection; Procedure: Breast Surgery; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Contrast Enhanced Digital Mammography; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Survey Administration; Procedure: Tissue Collection; Procedure: Ultrasound Imaging
- Arm II (Surgery + postoperative radiation therapy) (Experimental): Patients undergo SOC chemotherapy and SOC breast surgery followed by breast hypofractionated radiotherapy QD for a total of 5 fractions. Patients also undergo CT, MRI, PET, CEDM, and/or breast US throughout the study. Additionally, patients undergo a breast biopsy and may undergo optional blood sample collection and tissue collection on study.
  Interventions: Procedure: Biopsy of Breast; Procedure: Biospecimen Collection; Procedure: Breast Surgery; Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Contrast Enhanced Digital Mammography; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Survey Administration; Procedure: Tissue Collection; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Biopsy of Breast — Undergo breast biopsy
  Other Names: Breast Biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Breast Surgery — Undergo breast surgery
Drug: Chemotherapy — Receive SOC chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Contrast Enhanced Digital Mammography — Undergo CEDM
  Other Names: CEDM; Contrast Enhanced Spectral Mammography; Contrast-Enhanced Digital Mammography
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiotherapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Survey Administration — Ancillary studies
Procedure: Tissue Collection — Undergo tissue collection
  Other Names: Tissue Bank; Tissue Repository; Tissue/Specimen Collection
Procedure: Ultrasound Imaging — Undergo ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This phase II trial studies how well hypofractionated radiotherapy before (preoperative) or after (postoperative) breast surgery works in treating patients with different types of non-metastatic (has not spread from original tumor site) breast cancer and to determine the outcomes and side effects of this treatment. Radiation therapy is considered an integral part of breast conserving therapy. Hypofractionated radiation therapy is a radiation treatment in which the total dose of radiation is divided into large doses and treatments are given less than once a day. This has been shown to be an effective treatment for breast cancer while reducing treatment time and decreasing side effects. Preoperative radiotherapy alone or concurrently with chemotherapy has also been tested with excellent results and with minimal toxicity. Preoperative radiation of the intact tumor with a hypofractionated regimen can potentially decrease toxicity by allowing the delivery of treatment to intact breast tissue. The potential advantages of preoperative radiation therapy include the delivery of radiation in the intact breast when radiation can be more effective as more oxygen can be available in the tissue. Furthermore, complications and cosmetic results are expected to be lower in pre-operative radiotherapy before surgery, as there have been no changes in blood supply to the breast. This lends to the possibility of using lower doses of radiotherapy to patients, and potentially better cancer associated clinical outcomes for our breast cancer patients. Undergoing hypofractionated radiation therapy before or after breast surgery may be safe and effective in treating patients with different types of non-metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the rate of grade (G)3 or higher radiation treatment related adverse events with the use of preoperative and postoperative radiation within the first 2-years for groups A-D.

CORRELATIVE AND EXPLORATORY OBJECTIVES:

I. Grade 3 wound complications and seroma infection between preop and postoperative radiation.

II. Locoregional control with or without surgery at 2-years in group D (Her2+). III. To evaluate radiographic complete response and near complete response. IV. To estimate the 5-year locoregional control, distant recurrence, invasive disease-free survival, cause-specific survival, and overall survival.

V. To evaluate patient-reported outcomes. VI. To evaluate clinical features, treatment technique, dose-volume parameters, histologic and genetic variants associated with adverse events, and fair and poor cosmetic outcomes or unplanned surgical intervention.

VII. Evaluate tumor mutation signatures before and after chemotherapy, radiation, and surgery, correlate tumor mutation signatures before and after radiation with pathologic information at the time of surgery.

VIII. To describe the pathologic changes seen in breast cancer patients with preoperative radiation.

IX. Evaluate circulating tumor deoxyribonucleic acid (DNA), tumor infiltrating lymphocytes, neo-epitopes, and peripheral blood mononuclear before and after chemotherapy, radiation, and surgery; correlate tumor mutation signatures before and after radiation with pathologic information at the time of surgery.

X. Group A-D: Determine the rate of implant/tissue expander failure after preop and postop radiation.

XI. Group A-C: To determine the pathologic complete response (pCR) rate and near pathologic rate with cellularity <10% after neoadjuvant chemotherapy and hypofractionated radiotherapy to the whole breast with nodal irradiation if indicated, based on the postsurgical specimen.

XII. Group D: Determine locoregional control with the use of preoperative radiation conformal radiation. It will be determined based on the number of patients with controlled locoregional disease at 6-months.

XIII. Group A-C: To determine true radiographic complete response based on post treatment positron emission tomography (PET) standardized uptake value (SUV) <2.5 or uptake < mediastinum.

XIV. Group A-C: To determine the pathologic complete response (pCR) rate and near pathologic rate with cellularity <10% after neoadjuvant chemotherapy and hypofractionated radiotherapy to the whole breast with nodal irradiation if indicated, based on the postsurgical specimen.

XV. Group E: To determine the rates of surgery for locoregional disease after RT at 2 and 5-years.

XVI. Group E: To determine the rates of persistent disease in the breast or regional lymphatics after RT at 2 and 5-years.

OUTLINE: Patients with low risk and high risk estrogen receptor (ER) positive disease, triple negative disease and HER2 positive disease without complete response are randomized to 1 of 2 arms. Patients with HER2 positive, complete response disease are assigned to arm I.

ARM I: Patients undergo standard of care (SOC) chemotherapy followed by breast hypofractionated radiotherapy once daily (QD) for a total of 5 fractions. Patients then undergo SOC breast surgery 10 weeks after radiation treatment. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET), contrast-enhanced digital mammography (CEDM), and/or breast ultrasound (US) throughout the study. Additionally, patients undergo a biopsy and may undergo optional blood sample collection and tissue collection on study.

ARM II: Patients undergo SOC chemotherapy and SOC breast surgery followed by breast hypofractionated radiotherapy QD for a total of 5 fractions. Patients also undergo CT, MRI, PET, CEDM, and/or breast US throughout the study. Additionally, patients undergo a biopsy and may undergo optional blood sample collection and tissue collection on study.

After completion of study treatment, patients are followed up at 16 weeks, 6 months, 12 months, 24 months, 36 months, 48 months and at 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of breast cancer
* Clinical stage T1-T4 N0-3 M0
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2
* Able to and provides Institutional Review Board (IRB)-approved study specific written informed consent
* Able to complete all mandatory tests listed in the trial
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Indications for radiotherapy for breast cancer

Exclusion Criteria:

* Medical contraindication to receipt of radiotherapy
* Severe active co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or providing informed consent in the judgment of the principal investigator
* Active systemic lupus or scleroderma
* Pregnancy
* Women of childbearing potential who are unwilling to employ adequate contraception
* Prior receipt of ipsilateral breast or chest wall radiation
* Recurrent breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2031-10-21 (Estimated); Study Completion 2034-10-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher radiation treatment (RT) related adverse events | From baseline to 2 years after treatment initiation
  Will compare grade 3 or higher RT related adverse events with the use of preoperative and postoperative (Arm 1 versus Arm 2) radiation. Will be defined as an increase in the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 to grade 3+ compared to pre-radiation therapy. The primary analysis will be to estimate the adverse event rate within 2 years, defined as the cumulative incidence of patients experiencing the previously defined adverse events at any time from start of RT over the number of patients that have started RT at 2 years from the start of radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E. Vargas, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States